CLINICAL TRIAL: NCT05217953
Title: A Single-centre, Randomised, Cross-over Design Efficacy Study to Assess the Effectiveness of App-based, Assisted Behavioural Change Techniques to Improve HbA1c Levels and Support Diabetes Self-management in Young Adults and Adolescents
Brief Title: Improving HbA1c Levels Through Behavioural Change of Diabetes Self-management Assisted by the LovedBy Mobile Application for Young Adults and Adolescents With Type 1 Diabetes
Acronym: LBY-T1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: LovedBy LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B01038
Record Dates: First submitted 2022-01-18; First posted 2022-02-01 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This study will recruit 40 participants suffering from type-1 diabetes, split across 2 groups, with 30 needed for statistical significance (10 extra to allow for dropouts). The participant will have their average HbA1c levels measured (lab based, CONTROL-1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): The CGM will be integrated with the users mobile handset and all relevant measures taken will be entered. Participant will be provided with a smart watch and this will also be integrated with the users smartphone.
  The user will then download and install the LovedBy mobile app. Once installed the user will set up an account and the account number will be recorded by the clinical research team to track the participant throughout the trial. The final step is to review the permissions of the mobile application and allow the mobile application to connect to the users handset
  Interventions: Device: LovedBy App
- Control-Group (No Intervention): The same measurements will be taken as with the test group but here no app will be provided to the participants in this group.

INTERVENTIONS:
Device: LovedBy App — The LovedBy solution aims to leverage modern technologies such as smartphones, continuous glucose monitors (CGM), and other smart wearables to assist young sufferers managing their condition. The LovedBy platform offers a mobile application which connects to the user's smart wearables and CGM to monitor data streams that have been linked to long term risk. The mobile application is then able to deliver personally relevant educational content to the user through numerous channels including private social media message
  Arms: Test Group

SUMMARY:
Young people (16-25) with type-1 diabetes have historically struggled with managing their condition. Typically, the average HbA1c levels are significantly higher and as such, the risk of long term complications tend to be far greater.

These sufferers tend to have better management of their condition as they grow older however, the evidence suggests this is too late and these sufferers will likely have some complications later in life. Current cost to the NHS for complications is ~£850 million and expected to rise to ~£1.3 billion in the next 10-15 years.

The LovedBy solution aims to leverage modern technologies such as smartphones, continuous glucose monitors (CGM), and other smart wearables to assist young sufferers managing their condition. The LovedBy platform offers a mobile application which connects to the user's smart wearables and CGM to monitor data streams that have been linked to long term risk. The mobile application is then able to deliver personally relevant educational content to the user through numerous channels including private social media messages.

The study will last 10 months, and the participants are required to download/install the mobile app, integrate their wearables and then simply continue as normal with regular clinical meetings. Participants will be between 16-25 years and comply with the inclusion criteria set out in the protocol.

DETAILED DESCRIPTION:
This study will recruit 40 participants suffering from type-1 diabetes, split across 2 groups, with 30 needed for statistical significance (10 extra to allow for dropouts). The participant will have their average HbA1c levels measured (lab based, CONTROL-1). While the participants are participating in the trial, they will receive relevant educational content based on areas of management they are struggling with. The analysis that decides this is automated by the system which explores whether the particular criteria have been met for each educational pieces.

At the end of the study we will be able to compare whether the primary outcome has been met by comparing a final average HbA1c measure to CONTROL-1. Secondary outcomes can be evaluated using the sensor HbA1c recordings.

The entire study can be summarised as a reference to a reduction in long term risk and cost saving to the NHS.

Participant Journey

Pre-Trial (Visit 1):

1-3 hours 2-4 weeks before study starts Firstly, the patient will be sent all relevant study documents after which there is the recruitment call where the study will be described in detail. All risks will be discussed here and made clear. The data policies and management of data will also be described here. The patient will be able to ask any questions they wish to do so at this point.

If the patient is willing to participate in the trial, consent will be obtained after the they have had adequate time to reflect on the study.

Once consent has been obtained, the participant will be able to undergo lab HbA1c sampling. The participant will also undertake a questionnaire (Diabetes Distress Scale). The questionnaire will be undertaken at intervals between the other tasks during this visit.

Trial (Visit-2):

1-2 hours Study starts The clinical research team (CRT) will collect various measures such as weight, height blood pressure, body fat etc.and also ensure the users CGM is set up correctly.

Test-Group: The CGM will be integrated with the users mobile handset and all relevant measures taken will be entered. Participant will be provided with a smart watch and this will also be integrated with the users smartphone.

The user will then download and install the LovedBy mobile app. Once installed the user will set up an account and the account number will be recorded by the clinical research team to track the participant throughout the trial. The final step is to review the permissions of the mobile application and allow the mobile application to connect to the users handset. Control-Group: The same measurements will be taken as with the test group but here no app will be provided to the participants in this group.

Trial (Visit-3):

1-2 hours 8-weeks since last visit Test-Group: Participants of this group will undergo an interview with clinical research team. They will discuss events that were identified by the LovedBy platform. The CRT will also update the measures taken in the previous visit. The participant will also be asked to partake in a semi-structured interview to asses phycological efficacy.

Control-Group: This group will not undergo an interview.

Trial (Visit-4):

1-2 hours 8-weeks since last visit All participants will end the first arm of the study with lab HbA1c recorded. They will then proceed with a 4-week washout period. After which they will cross-over to begin the second arm of the study.

Trial (Visit-5):

1-2 hours 4-weeks since last visit This visit will be identical to Visit-2 but the Test-Group and Control-Group will switch over.

Trial (Visit-6):

1-2 hours 8-weeks since last visit This visit will be identical to Visit-3 where only the Test-Group will be interviewed.

Trial (Visit-7):

1-2 hours 8-weeks since last visit All participant will undergo a lab HbA1c sampling. The participant will undergo an exit interview regarding their experience with and without the LovedBy app. During this exit interview all LovedBy resources provided to the user such as smartwatches, CGM and applications will be handed back and/or removed from the user's device. The interview will aim to better capture the qualitative efficacy of the platform. It will be analysed to identify areas of design improvements that can be made on the user interface and content pieces.

Study Complete (Correspondence):

The participants will be provided the results of the study electronically

ELIGIBILITY:
Inclusion Criteria:

- 1. Age between 16 - 25. 2. Type 1 diabetes, as defined by World Health Organisation (WHO) for at least 1 year or is confirmed C-peptide negative. 3. HbA1c between 7.5 - 14.0% based on analysis from local laboratory or equivalent within 3 months of enrolment.

4. Has an Apple smartphone compatible with Dexcom G6. 5. Willingness to download the LovedBy app on their smartphone. 6. Willingness to wear an apple smartwatch. 7. Willingness to wear a Dexcom CGM. 8. Literate in English.

Exclusion Criteria:

* 1. Non-type 1 diabetes mellitus including those secondary to chronic disease. 2. Biphasic insulin MDI pen users. 3. Any other physical or psychological disease is likely to interfere with the normal conduct of the study.

  4. Untreated coeliac disease or hypothyroidism. 5. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids, Metformin, SGLT2 inhibitors, GLP-1 agonists, non-selective beta-blockers, MAO inhibitors etc.

  6. Medically documented allergy towards the adhesive (glue) of plasters or unable to tolerate tape adhesive in the area of sensor placement. 7. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin disease) located at places of the body, which could potentially be used for localisation of the glucose sensor. 8. Lack of reliable telephone facility for contact. 9. Known or suspected allergy against insulin. 10. Severe visual impairment. 11. Severe hearing impairment. 12. Not proficient in English. 13. Pregnancy, or planning for pregnancy.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-02-02 (Estimated); Study Completion 2024-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 4 months
  primary objective is to assess change in HbA1c change at 4 months following use of the LovedBy digital solution and 4 months without the the LovedBy app. (Lab based measures.)

SECONDARY OUTCOMES:
Time spent below target glucose (3.9 mmol/l) | 10 months
  Time spent below target glucose (3.9 mmol/l)
Time spent above target glucose (10.0 mmol/l) | 10 months
  Time spent above target glucose (10.0 mmol/l)
Average, standard deviation, and coefficient of variation of glucose levels | 10 months
  Average, standard deviation, and coefficient of variation of glucose levels
The time with glucose levels in hypoglycaemia at <3.5 mmol/l and <2.8 mmol/l | 10 months
  The time with glucose levels in hypoglycaemia at <3.5 mmol/l and <2.8 mmol/l
The time with glucose levels in significant hyperglycaemia (>16.7 mmol/l) | 10 months
  The time with glucose levels in significant hyperglycaemia (>16.7 mmol/l)
Total, basal and bolus insulin dose | 10 months
  Total, basal and bolus insulin dose
AUC of glucose below 3.5 mmol/l | 10 months
  AUC of glucose below 3.5 mmol/l

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No